CLINICAL TRIAL: NCT03372798
Title: INtra-procedural ultraSound Imaging for DEtermination of Atrial Wall Thickness and Acute Tissue Changes During Isolation of the Pulmonary Veins
Brief Title: INtra-procedural ultraSound Imaging During Pulmonary Veins Isolation
Acronym: INSIDEPVs
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Tim Betts MD MBChB FRCP, Principal Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 12163-SPON
Record Dates: First submitted 2017-03-22; First posted 2017-12-14 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Atrial Fibrillation
Keywords: catheter ablation; intraprocedural left atrial wall thickness imaging
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ICE/IVUS imaging during atrial fibrillation ablation — Intravascular ultrasound imaging of the left atrial wall thickness with ICE/IVUS during atrial fibrillation ablation

SUMMARY:
One of the biggest limitations of the currently used percutaneous techniques for Pulmonary Vein Isolation (PVI) in the setting of atrial fibrillation ablation is the lack of real-time information about the left atrial (LA) wall thickness and about its acute changes during energy delivery for ablation. This makes difficult to predict the achievement of transmural lesions, to identify the possible causes of ablation failure and also to avoid the occurrence of perforation and/or other collateral damage.

Computed tomography (CT) is a reliable technique for measurement of the LA wall thickness but it cannot be used during the ablation procedure and its extensive use is limited by the need of ionizing radiation. Preliminary data from animal studies support the accuracy of real-time ultrasound imaging modalities such as intracardiac echocardiography (ICE) or Intravascular Ultrasound (IVUS) imaging for measurement of LA wall thickness and monitoring of its acute changes related to catheter ablation.

The pilot study INSIDE PVs has been primarily designed to evaluate the feasibility and accuracy of intravascular imaging techniques for real-time imaging of the LA wall thickness during AF ablation.

DETAILED DESCRIPTION:
Patients scheduled for their first pulmonary vein (PV) isolation ablation for symptomatic, drug-refractory paroxysmal atrial fibrillation (AF), will be considered for inclusion in the study.

Potential subjects will initially be approached some weeks before their ablation procedure, in order to give the patients enough time to consider the information, to ask questions to the Investigator, their general practitioner (GP) or other independent parties to decide whether they wish to participate in the study or not.

For those interested in participation, a baseline assessment will be arranged to coincide with their standard pre-admission visit, for informed consent, screening and eligibility assessment. Moreover, a pre-operative imaging assessment with a cardiac computed tomography (CT) scan will be performed to define the left atrial (LA) and PV anatomy and to measure the baseline LA wall thickness and PVs ostial diameters.

All AF ablation procedures will be performed in a standard fashion by using radiofrequency (RF) energy, cryo-balloon or laser balloon ablation under general anaesthesia and with continuous oesophageal temperature monitoring. Ultrasound imaging by IVUS (Visions PV .018, 20 MHz digital probe, Volcano Corp) or ICE (Ultra ICE (9 MHz rotational transducer, Boston Scientific) will be performed at sites corresponding with the PV/LA junction at the beginning and the end of the procedure in order to measure acute changes in LA wall thickness and PV ostial diameters.

The cardiac CT will be repeated within 24 hours post-procedure. After the procedure, a pre-discharge review and a telephone follow-up at 1 week will be performed to identify any early and late complications related to the procedure.

A total of 14 patients will finally be enrolled in the study. The end of the study for each patient will be the date of the telephone follow-up 1 week after the procedure.

For each patient the pre-procedural and post-procedural CT measurements of LA wall thickness and PVs ostial diameters will be compared with the corresponding IVUS or ICE measurements.

ELIGIBILITY:
* Inclusion Criteria

  * Males older than 40 years or females older than 40 and sterile or in post-menopausal age;
  * willing and able to give informed consent for participation in the study;
  * history of symptomatic and drug-refractory paroxysmal atrial fibrillation (AF);
  * planned AF ablation on a clinical basis.
* Exclusion Criteria

  * age less than 40 years and more than 80 years;
  * pregnancy, trying for a baby or breast feeding;
  * any other significant disease or disorder which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study;
  * documented allergy to iodinated contrast medium;
  * renal insufficiency (eGFR<30);
  * weight exceeding the maximum load of the scanner (250kg).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective atrial fibrillation (AF) ablation in view of a history of symptomatic and drug-refractory paroxysmal AF.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Betts, MD, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kowalski M, Grimes MM, Perez FJ, Kenigsberg DN, Koneru J, Kasirajan V, Wood MA, Ellenbogen KA. Histopathologic characterization of chronic radiofrequency ablation lesions for pulmonary vein isolation. J Am Coll Cardiol. 2012 Mar 6;59(10):930-8. doi: 10.1016/j.jacc.2011.09.076. PMID 22381429
- [Background] Schwartzman D, Ren JF, Devine WA, Callans DJ. Cardiac swelling associated with linear radiofrequency ablation in the atrium. J Interv Card Electrophysiol. 2001 Jun;5(2):159-66. doi: 10.1023/a:1011477408021. PMID 11342752
- [Background] Weerasooriya R, Jais P, Sanders P, Scavee C, Hsu LF, Hocini M, Clementy J, Haissaguerre M. Images in cardiovascular medicine. Early appearance of an edematous tissue reaction during left atrial linear ablation using intracardiac echo imaging. Circulation. 2003 Sep 16;108(11):e80. doi: 10.1161/01.CIR.0000083530.08597.B5. No abstract available. PMID 12975247
- [Background] Khairy P, Dubuc M. Transcatheter cryoablation part I: preclinical experience. Pacing Clin Electrophysiol. 2008 Jan;31(1):112-20. doi: 10.1111/j.1540-8159.2007.00934.x. No abstract available. PMID 18181919
- [Background] Gage AA, Baust J. Mechanisms of tissue injury in cryosurgery. Cryobiology. 1998 Nov;37(3):171-86. doi: 10.1006/cryo.1998.2115. PMID 9787063
- [Background] Khairy P, Chauvet P, Lehmann J, Lambert J, Macle L, Tanguay JF, Sirois MG, Santoianni D, Dubuc M. Lower incidence of thrombus formation with cryoenergy versus radiofrequency catheter ablation. Circulation. 2003 Apr 22;107(15):2045-50. doi: 10.1161/01.CIR.0000058706.82623.A1. Epub 2003 Mar 31. PMID 12668527
- [Background] Reddy VY, Neuzil P, Themistoclakis S, Danik SB, Bonso A, Rossillo A, Raviele A, Schweikert R, Ernst S, Kuck KH, Natale A. Visually-guided balloon catheter ablation of atrial fibrillation: experimental feasibility and first-in-human multicenter clinical outcome. Circulation. 2009 Jul 7;120(1):12-20. doi: 10.1161/CIRCULATIONAHA.108.840587. Epub 2009 Jun 22. PMID 19546385
- [Background] Hall B, Jeevanantham V, Simon R, Filippone J, Vorobiof G, Daubert J. Variation in left atrial transmural wall thickness at sites commonly targeted for ablation of atrial fibrillation. J Interv Card Electrophysiol. 2006 Nov;17(2):127-32. doi: 10.1007/s10840-006-9052-2. Epub 2007 Jan 17. PMID 17226084
- [Background] Okada T, Yamada T, Murakami Y, Yoshida N, Ninomiya Y, Shimizu T, Toyama J, Yoshida Y, Ito T, Tsuboi N, Kondo T, Inden Y, Hirai M, Murohara T. Prevalence and severity of left atrial edema detected by electron beam tomography early after pulmonary vein ablation. J Am Coll Cardiol. 2007 Apr 3;49(13):1436-42. doi: 10.1016/j.jacc.2006.10.076. Epub 2007 Mar 21. PMID 17397672
- [Background] Granier M, Winum PF, Granier M, Liaud P, Cayla G, Messner P, Pasquie JL, Schuster I. Real-time atrial wall imaging during radiofrequency ablation in a porcine model. Heart Rhythm. 2015 Aug;12(8):1827-35. doi: 10.1016/j.hrthm.2015.04.012. Epub 2015 Apr 8. PMID 25863159
- [Background] Ren JF, Callans DJ, Schwartzman D, Michele JJ, Marchlinski FE. Changes in local wall thickness correlate with pathologic lesion size following radiofrequency catheter ablation: an intracardiac echocardiographic imaging study. Echocardiography. 2001 Aug;18(6):503-7. doi: 10.1046/j.1540-8175.2001.00503.x. PMID 11567596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment performed from November 2016 to October 2017 in Cardiology Outpatient Clinic.
  A total of 14 patients enrolled. 2 patients had incomplete datasets so 12 patients available for analysis.
Pre-assignment Details: Two recruited patients were not included in the data analysis because of
  * no intravascular ultrasound imaging available due to technical issue in 1 patient;
  * no post-operative CT scan performed by 1 patient.
Groups:
- Intracardiac Echo (ICE) Imaging: Pulmonary vein imaging performed during atrial fibrillation ablation with ICE
- Intravascular Ultrasound (IVUS) Imaging: Pulmonary vein imaging performed during atrial fibrillation ablation with IVUS
Period: Overall Study
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
Started | 8 | 6
Completed | 7 | 5
Not Completed | 1 | 1
Not completed — Patient not attending post-procedural CT scan | 1 | 0
Not completed — Failure of imaging probe | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11) | 63 (9) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 4 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 7 | 5 | 12
Ablation modality for Pulmonary Vein Isolation [Count of Participants; unit: Participants]
  Radiofrequency energy | 3 | 2 | 5
  Cryoenergy | 2 | 2 | 4
  Laser energy | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Left Atrial (LA) Wall Thickness on ICE/IVUS Frames
Description: Left atrial wall thickness at the PV ostia, measured as Wall Thickness Index % = [(vessel area - lumen area)/vessel area] x 100
Time Frame: Day 1
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
Number analyzed (Participants) | 7 | 5
percentage
  Pre-ablation | 22.18 [16.4 to 29.1] | 23.15 [20.8 to 27.8]
  Post-ablation | 27.04 [20.6 to 34.4] | 27.09 [22.8 to 32.3]

2. Primary Outcome: Measurement of LA Wall Thickness on CT Scans
Description: as for outcome 1
Time Frame: 1 day
Population: The analysis was not possible as the CT images were inadvertently deleted before any analysis was performed.
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Time Required for ICE/IVUS for Real Time Imaging of the Left Atrial (LA) Wall Thickness During AF Ablation
Description: Mean time required to image the left atrium for measurement of left atrial wall thickness with intracardiac echo (ICE) or with intravascular ultrasound (IVUS)
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
Number analyzed (Participants) | 7 | 5
minutes | 24.8 (3.4) | 25 (3.5)

4. Secondary Outcome: Number of ICE/IVUS Cases of Good Quality
Description: Number of intracardiac echo (ICE) cases and number of intravascular ultrasound (IVUS) cases of good quality, allowing a precise measurement of the left atrial (LA) wall thickness The imaging quality of each PV cross-section was defined as good quality if the vessel contour was visible in all 4 quadrants.
Time Frame: Day 1
Measure: Count of Units; unit: Pulmonary Vein cross-sections
Units Other Than Participants: Pulmonary Vein cross-sections
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
Number analyzed (Participants) | 7 | 5
Number analyzed (Pulmonary Vein cross-sections) | 28 | 20
Pulmonary Vein cross-sections | 24 | 0

ADVERSE EVENTS:
Time Frame: Day of catheter ablation procedure and one week after the procedure
Arm/Group | Intracardiac Echo (ICE) Imaging | Intravascular Ultrasound (IVUS) Imaging
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT03372798/Prot_SAP_000.pdf